CLINICAL TRIAL: NCT07182760
Title: Clinicopathologic Significance of Splenomegally in Adult Patients With Isolated Thrombocytopenia
Brief Title: Ultrasound to Detect Splenomegally in Patients With Isolated Thrombocytopenia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karim Ashraf hussein youssef, Resident in Internal Medicine Department in Assiut University Hospitals, Assiut University
Other Study IDs: S.I.TH
Record Dates: First submitted 2025-09-03; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Primary Immune Thrombocytopenic Purpura; Amegakaryocytic Aplasia; Unilineage Myelodysplastic Syndrome ( Megakaryocyte Dysplasia); Lymphoproliferative Disorder With Secondary ITP; Autoimmune Diseases With Secondary ITP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1a patients with isolated thrombocytopenia and splenomegaly: Group 1b patients with isolated thrombocytopenia without splenomegaly.
- Group 1b patients with isolated thrombocytopenia without splenomegaly.: Group 1b patients with isolated thrombocytopenia without splenomegaly.
- Group 2 healthy volunteers.

SUMMARY:
Investigate prevalence of splenomegally in patients with isolated thrombocytopenia.

Asess effect of splenomegally in clinical picture ,Complication, treatment response and disease outcome To explain possible causes of splenomegally in patients with isolated thrombocytopenia

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years admitted with isolated thrombocytopenia due to primary Immune thrombocytopenic purpura amegakaryocytic aplasia Unilineage myelodysplastic syndrome ( megakaryocyte dysplasia) lymphoproliferative disorder with secondary ITP autoimmune diseases with secondary ITP Willingness to participate in the study Admitted patients or those who follow at hematology outpatients clinic

Exclusion Criteria:

EDTA induced pseudothrombocytopenia Platelet satellitism Drug induced thrombocytopenia Heparin induced thrombocytopenia / thrombosis syndrome post transfusion purpura Disseminated intravascular coagulopathy patients less than 18 years old patients with bicytopenia or pancytopenia Pregnancy

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with isolated thrombocytopenia between 18 years to 65years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Investigate prevalence of splenomegally in patients with isolated thrombocytopenia. Asess effect of splenomegally in clinical picture ,Complication, treatment response and disease outcome | Baseline
  1. How many patients with isolated thrombocytopenia present with splenomegaly
  2. Do patients with splenomegaly experience different complications compared to those without splenic enlargement
  3. Is there a difference in treatment response between patients presenting with splenomegaly and those without splenic involvement

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Achterbergh R, Vermeer HJ, Curtis BR, Porcelijn L, Aster RH, Deenik W, Daemen-Gubbels C. Thrombocytopenia in a nutshell. Lancet. 2012 Feb 25;379(9817):776. doi: 10.1016/S0140-6736(11)61643-7. No abstract available. PMID 22364760
- [Background] Arnold J, Ouwehand WH, Smith GA, Cohen H. A young woman with petechiae. Lancet. 1998 Aug 22;352(9128):618. doi: 10.1016/s0140-6736(98)05194-0. No abstract available. PMID 9746024
- [Background] LAVY R. THROMBOCYTOPENIC PURPURA DUE TO LUPINUS TERMIS BEAN. J Allergy. 1964 Sep-Oct;35:386-9. doi: 10.1016/0021-8707(64)90065-6. No abstract available. PMID 14216353
- [Background] Kam T, Alexander M. Drug-induced immune thrombocytopenia. J Pharm Pract. 2014 Oct;27(5):430-9. doi: 10.1177/0897190014546099. Epub 2014 Aug 17. PMID 25134884